CLINICAL TRIAL: NCT05461508
Title: Study on the Effect of Fucoidan Combined With the Eradication Program Containing Vonoprazan on H.Pylori Eradication Rate and Gastrointestinal Flora.
Brief Title: Fucoidan Assisted Eradication of Helicobacter Pylori
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220518-02-KS-01
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Helicobacter Pylori Infection; Intestinal Bacteria Flora Disturbance
Keywords: Helicobacter Pylori Infection; Eradication treatment; Amoxicillin; vonoprazan; Fucoidan; Intestinal flora
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; fucoidan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin combined with vonoprazan (Active Comparator): The subjects will be given 20mg vonoprazan twice a day and 1000mg amoxicillin three times a day. These two drugs were taken continuously for 14 days
  Interventions: Other: Amoxicillin combined with vonoprazan
- Amoxicillin combined with vonoprazan and fucoidan (Experimental): The subjects will be given 20mg vonoprazan twice a day, 1000mg amoxicillin three times a day and fucoidan 1000mg twice a day. These three drugs were taken continuously for 14 days.
  Interventions: Biological: Amoxicillin combined with vonoprazan and fucoidan

INTERVENTIONS:
Biological: Amoxicillin combined with vonoprazan and fucoidan — Fucoidan was used in combination with amoxicillin and vonoprazan. The purpose of this study was to explore the effect of fucoidan on the eradication rate of Helicobacter pylori and the intestinal flora of subjects.
  Arms: Amoxicillin combined with vonoprazan and fucoidan
Other: Amoxicillin combined with vonoprazan — Amoxicillin and vonoprazan were used as the study control group
  Arms: Amoxicillin combined with vonoprazan

SUMMARY:
The purpose of this study is to investigate whether the eradication rate of H.pylori will be improved when adding fucoidan to the duplex scheme combination of amoxicillin and vonoprazan, and to explore the effect of fucoidan on gastrointestinal flora of patients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirement will be included in this simultaneous blind test. A total of 60 patients with HP infection were enrolled in this study. All patients were randomly divided into two groups according to the ratio of 1:1. Group A was given vonoprazan 20mg bid, amoxicillin 1000mg TID, fucoidan 1000mg bid for 14 consecutive days; Group B was given vonoprazan 20mg bid and amoxicillin 1000mg TID for 14 days. On the 10th and 14th days of treatment, the researchers will follow up the patients' adverse reactions and medication compliance. The feces of the subjects were collected one day before the treatment, and on the 14th and 44th days after the treatment; After 4 weeks of drug withdrawal, all subjects will be reexamined with 13C-UBT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Patients diagnosed as HP positive;
3. Patients who have not received HP eradication treatment in the past, or who have failed in the early eradication but have not received eradication treatment within half a year;
4. Voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

1. Allergic to the study drug (penicillin allergy, etc.);
2. Patients with chronic gastritis and peptic ulcer;
3. Patients who have received HP eradication treatment within half a year;
4. Antibiotics and bismuth agents were used 4 weeks before the start of the study treatment, and histamine H2 receptor antagonists or PPIs were used 2 weeks before the start of the study treatment;
5. Use adrenocortical hormones, non steroidal anti-inflammatory drugs or anticoagulants;
6. History of esophageal or gastric surgery;
7. Pregnant and lactating women;
8. Suffering from serious accompanying diseases, such as liver disease, cardiovascular disease, lung disease, kidney disease;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
compare eradication rates of the two groups by 13C-UBT | 6 weeks
  Compare the eradication rate of Helicobacter pylori between the fucoidan containing group and the fucoidan free group
Analysis of intestinal flora difference before and after eradication using 16s rRNA sequencing | 6 weeks
  Analyze and compare the early and long-term changes of intestinal flora before and after eradication. Explore the effect of fucoidan on intestinal flora of patients receiving eradication treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China